CLINICAL TRIAL: NCT03255525
Title: Deep Friction Massage Effects on Analgesia of the Asymptomatic Patellar Tendon
Brief Title: Deep Friction Massage Effects: Asymptomatic
Acronym: DFM_Asymp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cooperativa de Ensino Superior, Politécnico e Universitário (Other)
Responsible Party: Principal Investigator, Maria Paço, PhD, Clinical research, Cooperativa de Ensino Superior, Politécnico e Universitário
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DFM_1
Record Dates: First submitted 2017-08-18; First posted 2017-08-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Deep Friction Massage

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Deep friction massage P50 (Active Comparator): In this group it was applied a pressure previously found to be the mean pressure applied by physiotherapists during deep friction massage.
  Interventions: Other: Deep friction massage P50
- Deep friction massage P25 (Experimental): In this group it was applied the percentile 25, of the pressure previously found to be the mean pressure applied by physiotherapists during deep friction massage.
  Interventions: Other: Deep friction massage P25
- Deep friction massage P75 (Experimental): In this group it was applied the percentile 75, of the pressure previously found to be the mean pressure applied by physiotherapists during deep friction massage.
  Interventions: Other: Deep friction massage P75

INTERVENTIONS:
Other: Deep friction massage P50 — Deep friction massage as described by Dr. James Cyriax, applied with the mean pressure (P50)
  Arms: Deep friction massage P50
Other: Deep friction massage P25 — Deep friction massage as described by Dr. James Cyriax, applied with the percentile 25 of the mean pressure (P25)
  Arms: Deep friction massage P25
Other: Deep friction massage P75 — Deep friction massage as described by Dr. James Cyriax, applied with the percentile 75 of the mean pressure (P75)
  Arms: Deep friction massage P75

SUMMARY:
Despite DFM being a widely-used technique and the empirical grounding regarding the importance of the pressure applied, there is no study characterizing the pressure applied during DFM, remaining it a discretion of the physiotherapist. Additionally, it is not known how the amount of pressure applied may influence pain mechanisms and, consequently how it affects the time needed promote an analgesic response.

Having this, our general objective is to establish a dose-response relationship between the pressure applied during DFM and time of onset of analgesia, in the asymptomatic patellar tendon.

ELIGIBILITY:
Inclusion Criteria:

* the participants should have an asymptomatic patellar tendon

Exclusion Criteria:

* history of previous injury of the lower limbs;
* intake of medication that could interfere with pain mechanisms;
* presence of any factors or conditions that could interfere with the tendinous tissue as well as with the awareness and sensibility to pain.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

PRIMARY OUTCOMES:
Time until analgesia | 10 minutes
  Self reported sensation of analgesia, controlled by a chronometer

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Paço, PhD, Principal Investigator — Cooperativa Ensino Superior Politécnico e Universitário
Locations (1):
- Cooperativa Ensino Superior Politécnico e Universitário, Gandra, Paredes, Portugal

IPD SHARING:
Plan to Share IPD: No